CLINICAL TRIAL: NCT04991441
Title: Impact of a Low-Sodium Meal Feeding Protocol on Interdialytic Weight Gain and Markers of Cardiovascular Health in Hemodialysis Patients
Brief Title: Dietary Sodium-Restriction (DIS) and Renal Meals (RM) for Hemodialysis (HD)(DISaRM-HD)
Acronym: DISaRM-HD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19507
Record Dates: First submitted 2021-03-30; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2020-12

CONDITIONS: Kidney Failure, Chronic; Dietary Modification
Keywords: Chronic Kidney Disease; Hemodialysis; Sodium Restriction
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Observational control followed by dietary intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Participants will follow their usual or normal diet for 5 months (CON) followed by an Controlled Dietary Sodium Restriction (INT) diet for 2 months. During the sodium restricted diet, participants will be provided with 2 meals and snacks daily, for 30 days (Month 5 - days 1-30) and 1 meal and snacks daily, for 30 days (Month 6 - days 31-60). These meals should meet the National Kidney Foundation's Kidney Disease Outcomes Quality Initiative (KDQOI) guidelines for energy and protein (30-35 kcal/kg & 1.2 g/kg) as well as low phosphorus, potassium, and sodium. The meals are formulated to less than 600-800 mg sodium each (<2,000g/day) and will be ordered and delivered through momsmeals.com
  Interventions: Dietary Supplement: Controlled Dietary Sodium Restriction; Dietary Supplement: Control Diet & Controlled Dietary Sodium Restriction
- Intervention (Experimental): Participants will be provided with 2 meals and snacks daily, for 30 days (days 1-30) and 1 meal and snacks daily, for 30 days (days 31-60). These meals should meet KDQOI guidelines for energy and protein (30-35 kcal/kg & 1.2 g/kg) as well as low phosphorus, potassium, and sodium. The meals are formulated to less than 600-800 mg sodium each (<2,000g/day) and will be ordered and delivered through momsmeals.com
  Interventions: Dietary Supplement: Control Diet & Controlled Dietary Sodium Restriction

INTERVENTIONS:
Dietary Supplement: Controlled Dietary Sodium Restriction — Participants will be provided with 2 meals and snacks daily, for 30 days (days 1-30) and 1 meal and snacks daily, for 30 days (days 31-60). These meals should meet KDQOI guidelines for energy and protein (30-35 kcal/kg & 1.2 g/kg) as well as low phosphorus, potassium, and sodium. The meals are formulated to less than 600-800 mg sodium each (<2,000g/day) and will be ordered and delivered through momsmeals.com
  Other Names: INT
  Arms: Control
Dietary Supplement: Control Diet & Controlled Dietary Sodium Restriction — Participants will follow a Observational Control Diet (CON) diet (Months 1-5) followed by an Controlled Dietary Sodium Restriction (INT) diet (Months 6-7).
  Other Names: CON

SUMMARY:
Chronic volume overload (VO) is a primary factor responsible for the excessive cardiovascular morbidity and mortality in hemodialysis (HD) patients. VO is caused in part by excessive fluid intake that is secondary to the consumption of a high salt diet. HD patients are often counselled to restrict their dietary sodium intake to help manage thirst and reduce their interdialytic weight gain (IDWG). However, data from recently published investigations demonstrate that dietary counseling alone may be ineffective. The objective of this randomized controlled trial is to determine if short-term feeding of low-sodium meals can "prime" changes in long-term nutrition behavior. It is hypothesized that feeding low-sodium meals for one month will significantly reduce IDWG and related outcomes, and continued dietary counseling and education support for 6 months will result in a sustained reduction in sodium intake upon patient resumption of meal responsibility. HD patients will be recruited and randomized to 2 groups: 1) Low-sodium meal feeding plus dietary counseling; or 2) a weight-list control group that will initially receive dietary counseling alone. IDWG will serve as the primary outcome with fluid volume overload, intradialytic hypotension, cramping, dietary sodium intake, sodium taste sensitivity and preference, and sodium self-efficacy evaluated at 1 and 6 months. This outcomes of this investigation will provide the first data on whether meal provision is an effective tool for dietary modeling and prolonged behavior change in HD patients.

DETAILED DESCRIPTION:
Chronic kidney disease patients with end-stage renal disease require regular hemodialysis (HD) therapy 3-4 days per week to filter their blood of toxins/waste and to remove excess fluid. HD therapy is essential for survival in patients with kidney failure, but the dialysis process is inefficient and does not remove all of the fluid and waste products that accumulate in patients since their last treatment. The inefficiency of dialysis, coupled with excessive dietary sodium and fluid intakes, results in a high prevalence of chronic volume overload (VO) and VO dependent hypertension (HTN). Both VO & HTN can have adverse effects on the heart and arteries, eventually lead to enlargement of the heart and cardiac dysfunction (1-3).

Dialysis care providers (doctors, dietitians, technicians) provide regular counseling for patients to reduce their dietary sodium and fluid intake, despite widespread non-adherence and the high prevalence of both VO and hypertension. Research interventions to increase dietary education and support behavior change have also demonstrated low efficacy in the dialysis patient population. Many barriers and factors contribute to excessive dietary sodium intakes and poor dietary adherence, thus is appears that current dietary education strategies may not be robust enough to change patient behaviors. However, a recent study in heart failure patients demonstrated that home-delivered meals represent a unique opportunity alter outpatient dietary practices. Patients with multiple comorbidities and numerous dietary behaviors, such as those on renal replacement therapy, may need additional support to establish and maintain dietary changes.

The purpose of this study is to compare dietary counseling with renal home meal delivery on clinical outcomes relating to both VO & HTN. This trial is a comparative-effectiveness mixed-models design. In this study, patients will be randomized to one of two study arms: 1) CON (7 months total) where patients receive usual care (eating their normal diet) for the first 5 months of the study. This will be followed by a 2-month period where they will receive home-delivered meals and additional dietary counseling to reduce sodium intake; OR 2) INT (5 months total), where patients will receive home-delivered meals plus additional dietary counseling for the first 2 months of the study, followed by 3 months of continued counseling. During the home-meal delivery periods, participants will be provided a low-sodium/renal diet that includes receiving 2 meals per day during their 1st month, and 1 meal per day during the 2nd month (month 6 and 7 for CON; and month 1 and 2 for INT). The meals will be delivered to the participant's homes each week by momsmeals.com.

We are also plan to collect sensory taste data to characterize patients on dialysis preferences for salt. It is possible that a low sodium diet may change these preferences, so that patients desire more low-sodium tasting food. This information would allow us to analyze how dialysis patients salt intake is associate with taste preference with salt and how this relates to clinical outcomes. The study outcomes include: clinical outcomes (hospitalizations, treatment efficiency), cardiovascular measures (blood pressure, cardiac output, and vascular resistance) and fluid/hydration status (total body water, extracellular fluid) using bioelectrical impedance.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to sign informed consent document and age 18 or greater.
2. High fluid gainer/excessive overloaded defined by: > 3.0 % of estimated-dry weight (EDW)
3. No upper or lower limb amputations. This criteria is necessary because the BIS device we are using is not able to provide accurate estimates of fluid status in participants with limb amputations.
4. No pacemakers
5. Willingness to consume intervention meals provided throughout the study.

Exclusion Criteria:

* not meeting above inclusion criteria 1 - 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessing Interdialytic weight gain (IDWG) using bioelectric impedance spectroscopy device (BIS) | Five months
  The research team will assess patients hydration status by using a non-invasive Cardiac System (NICaS) bioelectric impedance spectroscopy device (BIS) that will focus on noninvasive assessment and monitoring of cardiovascular, respiratory, and fluid parameters. The system provides real-time data on various parameters of a patient's cardiac and vascular functions. NICaS is a method of Impedance Cardiography (ICG) which utilizes dual impedance electrodes (about 3''x3''), placed on two limbs, preferably one on the wrist and the other on the contralateral ankle (any combination may work). NICaS measurements include the cardiac output and its derivatives, as well as an assessment of the left ventricular cardiac contractility. This device will be used to measure fluid retention between treatments.
Blood Pressure - markers of cardiovascular risk | Five months
  The research team will use an IntelliSense® Blood Pressure Monitor to measure blood pressure accurately prior to dialysis treatment in quiet conditions with participants sitting rested for approximately 10 minutes. This measurement will take less than 2 minutes total to complete. The systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) will be collected for this outcome.

SECONDARY OUTCOMES:
Dietary Recalls using ASA24 | Five months
  The research team will meet with each study participant to go over weekly nutrition education. Topics will include various activities such as reading a nutrition label, identifying 'high sodium' and 'low sodium' food content at grocery stores, introduction to 'low sodium' recipes, and cooking with alternative salt-free spices. In addition, the research team will use the Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool to assess diet recalls. The ASA24 is a web-based tool that enables multiple, automatically coded self-administered 24-hour recalls and/or multi- day food records also known as food diaries. The National Cancer Institute (NCI) provides ASA24 to the research community at no cost. Diet recalls will serve to document the change in sodium intake through the duration of the study. The sodium content (mg) of the food participants eat will be used for this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Wilund, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigative team will disseminate data from this study through publication in scientific journals, as well as at academic seminars and professional conferences and meetings in the fields of nutrition and Nephrology.
Time Frame: The investigative team will disseminate data from this study through publication in scientific journals, as well as at academic seminars and professional conferences and meetings in the fields of nutrition and Nephrology.
Access Criteria: The investigative team will disseminate data from this study through publication in scientific journals, as well as at academic seminars and professional conferences and meetings in the fields of nutrition and Nephrology.